CLINICAL TRIAL: NCT05494684
Title: Effectiveness of Multisensoral Nature-based Intervention in Hospitalized Children Aged 5 to 9 Years During Venous Blood Sampling: A Randomized Controlled Trial
Brief Title: Effectiveness of Multisensoral Nature-based Intervention in Hospitalized Children During Venous Blood Sampling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Saija Huhtala, Principal Investigator, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08072402
Record Dates: First submitted 2022-07-29; First posted 2022-08-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Fear; Pain; Satisfaction
Keywords: Children; Nature-based Intervention; Venipuncture
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomization of the children participating in the study will be carried out using the Stratified Block Randomization-on method, which allows randomization in two groups, according to age, as follows: group 1 (5-6 years old) and group 2 (7-9 years old). This is to ensure that the intervention and control groups have the same number of children of the same age and do not differ in their starting level. The randomization lists are made by a statistician.
Who Masked: Outcomes Assessor
Masking Description: The children blood sampling will be videotaped. The principal investigator videos the blood sampling, and then external observer assesses the child's anxiety (mYPAS=Modifield Yale preoperative anxiety scale) on video. The video camera is pre-installed in the blood sampling room and positioned so that it does not attract attention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Children and parents receive a multisensoral nature-based intervention during venous blood sampling.
  Interventions: Other: Multisensoral Nature-based Intervention
- Control Group (No Intervention): The control group receives the usual standard care during venous blood sampling

INTERVENTIONS:
Other: Multisensoral Nature-based Intervention — The intervention includes a multi-sensory nature experience using natural materials and a virtually created natural environment.
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial (RCT) study aims to evaluate the effectiveness of multisensoral nature-based intervention compare to standard care in relieving anxiety, fear and pain in hospitalized child aged 5 to 9 years and parent's anxiety and satisfaction during venous blood sampling. The assessment uses different measures to assess child's anxiety, fear, pain and parent's anxiety and satisfaction during venous blood sampling.

DETAILED DESCRIPTION:
The RCT study aims to evaluate the effectiveness of multisensoral nature-based intervention compare to standard care in relieving anxiety, fear and pain in hospitalized child aged 5 to 9 years and parent's anxiety and satisfaction during venous blood sampling. The intervention includes a multi-sensory nature experience using natural materials and a virtually created natural environment. The study will include children and parents in the intervention group (N=53, receiving the multisensoral nature-based intervention) and children and parents in the control group (N=53, receiving usual care). The children's blood sampling will be videotaped. The assessment uses different measures assess to child's anxiety (mYPAS = The modified Yale preoperative anxiety scale), child's fear (CFC = Children Fear Scale), child's pain (FAS = Facial Affective Scale), parent's anxiety (STAY-Y1 = The State-Trait Anxiety Inventory) and satisfaction (VAS = Visual Analogue Scale) during venous blood sampling. In addition, heart rate (HR) measurement are used to assess the child's anxiety, fear and pain. The data will be analysed using statistical methods.

ELIGIBILITY:
Inclusion Criteria:

1. The child is aged between 5 and 9 years old
2. The child has a long-term illness (such as diabetes or rheumatism)
3. The child has previous experience of venous blood sampling
4. The child's level of development is age-appropriate (such as, the child is cared for at home or in day care/day nursery or attends school in the same level as the other children)
5. Child and parent understand and speak the Finnish language

Exclusion Criteria:

1. The child has a diagnosis of abnormal neurological development (such as, a child has difficulty understanding spoken language or expressing emotions)
2. The child has chronic pain that has lasted more than 3 months and requires strong painkillers (opiates).
3. The child undergoes an examination or treatment during a check-up at the outpatient clinic that requires medical treatment similar to anesthesia
4. The child is taking a sedative medication.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety measured with mYPAS (the modifield Yale preoperative anxiety scale). An external observer assesses the child's anxiety before blood sampling on video. | Before blood sampling
  The mYPAS (modifield Yale preoperative anxiety scale) was developed for external observers to assess a child's anxiety before blood sampling and is suitable for measuring anxiety in children aged 2-16 years. The Modifield Yale preoperative scale measures the child's activity, voice, emotional expression and parental need (1-4/4, 1-6/6, 1-4/4, 1-4/4 points). Each item is scored separately and the total score is multiplied by 20. The lowest score for child anxiety is 1 and the highest score is 100. The scale has been tested for validity and relational validity (Kain X.N. et al. 1997).

SECONDARY OUTCOMES:
Fear measured with CFS (Children Fear Scale). Child and parent assessment of fear during blood sampling. | During blood sampling
  The Children Fear Scale (CFS) is a modified version of the anxiety scale (McKinley et al. 2004). The five-item, gender-neutral, visual face scale measures fear in children aged 5-10 years and can be used during blood sampling. Images are viewed from left to right, from non-fearful faces to very fearful faces (0-4 points). On the Children Fear Scale, unafraid faces score 0 points and very fearful faces score 4 points. The validity and relative validity of the scale have been tested (McMurtry et al. 2011).
Pain measured with FAS (Facial Affective Scale). Child and parent assessment of pain during blood sampling. | During blood sampling
  The Facial Affective Scale (FAS) (McGrath et al. 1996) measures the intensity of pain in children over 5 years of age and can be used during blood sampling. The Facial Affective Scale assesses a child's pain using nine facial images, presented in order from the happiest face (0.04 points) to the saddest face (0.97 points). A happy face (0.04 points) indicates no pain and a sad face (0.97 points) indicates very painful. The FAS score assesses the child's emotional or affective response to the experience of pain (Nguyen et al. 2010). The scale has been tested for validity and relative validity (Nilsson et al. 2014).
Parent's anxiety with STAI-Y1 (The State-Trait Anxiety Inventory). Parent self-assessment of own anxiety before blood sampling. | Before blood sampling
  The State-Trait Anxiety Inventory (STAI-Y1) measures an adult's anxiety, tension, fear and worry at the moment. The State-Trait Anxiety Inventory is a 4-point Likert scale (not at all anxious, number 1, somewhat anxious, number 2, moderately anxious, number 3, and very anxious, number 4) with 20 different questions. The State-Trait Anxiety Inventory STAI-Y1 measures situational anxiety (Copyright © 1983 by Charles D. Spielberger), in which the parent selects the number that best describes their own feelings at the moment. This study measures parent anxiety before blood sampling. The scale has been tested for validity and relational validity (Nilsson et al. 2014).
Parent's satisfaction with VAS (A Visual Analogue Scale). Parent self-assessment of own satisfaction after blood sampling. | After blood sampling
  The VAS (A Visual Analogue Scale) assesses parent satisfaction on a scale of 0-10 after a blood sampling, where 0 means not at all satisfied and 10 means very satisfied.The scale has been tested for validity and relational validity (Abu-Saad 1984).
Child's anxiety, fear and pain with physiological measures: Heart Rate (HR, beats per minute) during blood sampling. | During blood sampling
  The child's heart rate (HR, beats per minute) was measured during blood sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Saija Huhtala, Principal Investigator — Oulu University
Locations (1):
- Oulu Univeristy, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] McKinley S, Stein-Parbury J, Chehelnabi A, Lovas J. Assessment of anxiety in intensive care patients by using the Faces Anxiety Scale. Am J Crit Care. 2004 Mar;13(2):146-52. PMID 15043242
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307
- [Background] Nguyen TN, Nilsson S, Hellstrom AL, Bengtson A. Music therapy to reduce pain and anxiety in children with cancer undergoing lumbar puncture: a randomized clinical trial. J Pediatr Oncol Nurs. 2010 May-Jun;27(3):146-55. doi: 10.1177/1043454209355983. PMID 20386063
- [Background] Nilsson S, Finnstrom B, Morelius E, Forsner M. The facial affective scale as a predictor for pain unpleasantness when children undergo immunizations. Nurs Res Pract. 2014;2014:628198. doi: 10.1155/2014/628198. Epub 2014 Mar 5. PMID 24734174
- [Background] Abu-Saad H. Assessing children's responses to pain. Pain. 1984 Jun;19(2):163-71. doi: 10.1016/0304-3959(84)90836-4. PMID 6462728